CLINICAL TRIAL: NCT01939574
Title: An Open-label, Single Arm Study to Explore Whether Potential Image Biomarkers Correlate With Efficacy of Bevacizumab Combined With Conventional Therapy in Newly Diagnosed Glioblastoma
Brief Title: A Explore Study of Bevacizumab Combined With Conventional Therapy in Glioblastoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinming Yu, Professor, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML28676
Record Dates: First submitted 2013-09-02; First posted 2013-09-11 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Glioblastoma
Keywords: Glioblastoma; Potential Image Biomarkers; PFS; Bevacizumab; Conventional Therapy
MeSH Terms: conditions — Glioblastoma | interventions — Neoadjuvant Therapy; Radiotherapy; Temozolomide; Bevacizumab; Chemotherapy, Adjuvant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Chemoradiation & Adjuvant Therapy: (Experimental): * Concurrent chemoradiation Therapy:
    * Radiation therapy:2 Gy will be given daily 5 days per week for a total of 60 Gy over 6 weeks.
    * Temozolomide from day 1 of radiotherapy to the last day of radiation at a daily oral dose of 75 mg/m2 for a maximum of 49 days.
    * Bevacizumab will be administered intravenously on days 1 and 15 of each 28-day cycle,at the beginning of the 4th week of radiation. The dose will be 10 mg/kg.
  * Adjuvant Therapy:
    * Temozolomide once per day for 5 consecutive days of a cycle. The starting dose for the first cycle will be 150 mg/m2/day, with a single dose 200 mg/m2/day in subsequent cycles if no treatment-related adverse events> grade 2 are noted.
    * Bevacizumab will be administered intravenously on days 1 and 15 of each 28-day cycle. The dose will be 10 mg/kg.
  Interventions: Other: Chemoradiation Therapy; Other: Adjuvant Therapy

INTERVENTIONS:
Other: Chemoradiation Therapy — * Radiation therapy:For both intensity-modulated radiation therapy (IMRT) and three-dimensional conformal radiation therapy (3D-CRT) plans, one treatment of 2 Gy will be given daily 5 days per week for a total of 60 Gy over 6 weeks.
  * Temozolomide will be administered continuously from day 1 of radiotherapy to the last day of radiation at a daily oral dose of 75 mg/m2 for a maximum of 49 days.
  * Bevacizumab will be administered intravenously on days 1 and 15 of each 28-day cycle,at the beginning of the 4th week of radiation. The dose will be 10 mg/kg of actual body weight.
  Other Names: Radiation therapy; Temozolomide; Bevacizumab
Other: Adjuvant Therapy — * Temozolomide will be administered orally once per day for 5 consecutive days (days 1-5) of a 28-day cycle. The starting dose for the first cycle will be 150 mg/m2/day, with a single dose escalation to 200 mg/m2/day in subsequent cycles if no treatment-related adverse events> grade 2 are noted.
  * Bevacizumab will be administered intravenously on days 1 and 15 of each 28-day cycle. The dose will be 10 mg/kg of actual body weight.
  Other Names: Temozolomide; Bevacizumab

SUMMARY:
This is a single-center, open-label, single arm study to explore whether potential image biomarkers correlate with efficacy of bevacizumab combined with conventional therapy in newly diagnosed glioblastoma.

Despite the increase in therapies available, the median survival of patients with glioblastoma multiforme (GBM) remains less than 15 months.

The phase III pivotal study in newly diagnosed GBM also met its co-primary endpoint of progression-free survival (PFS) which further confirm the efficacy of bevacizumab in GBM.

Early predicting the efficacy of bevacizumab combined with conventional therapy in newly diagnosed glioblastoma could help us to identify the suitable patients to receive suitable treatment in GBM. Thus, characterizing the blood flow and blood volume in the tumor and their changes during therapy might provide information on vasculature growth or collapse,edema formation, tumor growth, and/or cell death(necrosis) .We decided to investigate whether the estimation of blood circulation in tumor, using MRI,PET could be used as a surrogate marker to predict the early response of GBM to bevacizumab.

Several previous studies have demonstrated that the relative cerebral blood volume (rCBV) correlated with the histologic grade of gliomas and investigated the prognostic value of the tumor CBV for survival.In current study, We hypothesized that, the temporal changes during anti-angiogenesis therapy in specific regions of high and low perfusion in glioblastoma might predict the efficacy of bevacizumab.Since there is no mature PET tracer directly image Vascular Endothelial Growth Factor (VEGF) in China,we use 18F-Galacto-arginine-glycine-aspartic acid (RGD)-- a new tracer for PET imaging of αvβ3 by testing Standardized uptake value mean (SUVmean),Standardized uptake value max (SUVmax) and tumor to non-tumor tissue ratios (T/NT) to indirectly reflect the VEGF expression. The integrin αvβ3 is an important receptor affecting tumor growth, local invasiveness, and metastatic potential. Specifically, αvβ3 is highly expressed on activated endothelial cells during angiogenesis.

Therefore, in the pilot study, we use dynamic contrast enhanced magnetic resonance imaging (DCE-MRI),dynamic susceptibility-contrast magnetic resonance imaging (DSC-MRI) and 18F-Galacto-RGD PET to explore the potential image biomarkers of bevacizumab used in newly diagnosed glioblastoma.

DETAILED DESCRIPTION:
20 patients with newly diagnosed histopathologically confirmed glioblastoma (WHO Grade IV) after surgery will be enrolled in the study. All of the patients will receive conventional concurrent chemoradiation and adjuvant temozolomide plus bevacizumab begin > 3 weeks and ≤ 5 weeks after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven newly diagnosis of glioblastoma (WHO grade IV)
* The tumor must have a supratentorial component
* The patient must have recovered from the effects of surgery, postoperative infection, and other complications before initial chemoradiation treatment
* Documentation of steroid doses within 14 days prior to initial chemoradiation treatment
* Karnofsky performance status ≥ 70;
* Age ≥ 18
* Adequate renal function,hepatic function
* Systolic blood pressure ≤ 160 mg Hg or diastolic pressure ≤ 90 mg Hg within 14 days prior to initial chemoradiation treatment
* Patient must provide study specific informed consent prior to study entry
* Women of childbearing potential and male participants must practice adequate contraception.
* For females of child-bearing potential, negative serum pregnancy test within 14 days prior to initial chemoradiation treatment

Exclusion Criteria:

* Cancer-Related Exclusion Criteria

  * Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥3 years
  * Recurrent or multifocal malignant gliomas
  * Metastases detected below the tentorium or beyond the cranial vault
  * Prior chemotherapy or radiosensitizers for cancers of the head and neck region; note that prior chemotherapy for a different cancer is allowable, except prior temozolomide or bevacizumab. Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment are not permitted.
  * Prior radiotherapy to the head or neck (except for T1 glottic cancer), resulting in overlap of radiation fields
* Haematologic, Biochemical, Organ Function and other general exclusion criteria

  * Unstable angina and/or congestive heart failure within the last 6 months
  * Transmural myocardial infarction within the last 6 months
  * Evidence of recent myocardial infarction or ischemia by the findings of S-T elevations of ≥ 2mm using the analysis of an EKG performed within 14 days of initial chemoradiation treatment
  * New York Heart Association grade II or greater congestive heart failure requiring hospitalization within 12 months prior to initial chemoradiation treatment
  * History of stroke, cerebral vascular accident (CVA) or transient ischemic attack within 6 months
  * Serious and inadequately controlled cardiac arrhythmia
  * Acute bacterial or fungal infection requiring intravenous antibiotics at the time of registration
  * Chronic obstructive pulmonary disease exacerbation or other respiratory illness requiring hospitalization or precluding study therapy at the time of initial chemoradiation treatment
  * Hepatic insufficiency resulting in clinical jaundice and/or coagulation defects; note, however,that laboratory tests for liver function and coagulation parameters are not required for entry into this protocol
  * Inability to undergo MRI (e.g., due to safety reasons,such as presence of a pacemaker) or PET
* Contradiction to Bevacizumab treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2013-08; Primary Completion 2016-06 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Correlation between image biomarker change and PFS | At Week 10 of the study
  PFS (evaluated by RANO criteria), defined as the interval from start of treatment to investigator-assessed progression or death, whichever occurs first or lost of follow-up.
  At Week 10 of the study (corresponding to 7 weeks after the commencement of bevacizumab therapy).

SECONDARY OUTCOMES:
To assess overall survival(OS) | Up to 106 weeks
  OS is the time interval from the start of treatment to death due to any reason or lost of follow-up.
To evaluate the overall response rate (ORR) | At baseline, on day 22, 70, 127, end of treatment and every 2 months of follow-up
  ORR is the number of responders (CR, PR) vs. the whole study population.Tumor response will be evaluated according to the Response Assessment in Neuro-Oncology (RANO) criteria.
To evaluate health-related quality of life | On day 1, 22, 71, end of treatment and every 2 months of follow-up
  European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core-30
To assess the safety profile | Up to 106 weeks
  Safety will be measured based on the NCI-Common Terminology Criteria for Adverse Events (NCI-CTCAE), v4.0

CONTACTS AND LOCATIONS:
Overall Officials: Jinming Yu, PhD, Study Chair — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided